CLINICAL TRIAL: NCT00851071
Title: Bakken Heart Brain Institute's "An Observational and Interventional Study of Anxiety Symptoms in the Implantable Cardioverter Defibrillator (ICD) Patient."
Brief Title: Interventional Study of Anxiety Symptoms in the Implantable Cardioverter Defibrillator (ICD) Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Mina Chung, MD, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB# 08-913
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Anxiety
Keywords: Anxiety; Implantable Cardioverter Defibrillator (ICD); Defibrillators, Implantable
MeSH Terms: conditions — Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy (Active Comparator): Three individual 45 minute cognitive behavioral therapy sessions over a 3 month period
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Usual Care Arm (No Intervention): The Usual Care Arm will be the control arm. These patients will not be scheduled with any CBT sessions.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Three 45 minute CBT sessions scheduled over a 3 month period.
  Arms: Cognitive Behavioral Therapy

SUMMARY:
This study will compare the effectiveness that Cognitive Behavioral Therapy has on decreasing the amount of anxiety, as well as the number of inappropriate firings that a patient with an ICD may experience.

DETAILED DESCRIPTION:
This study is an interventional study of patients with ICDs followed in the Cleveland Clinic Device Clinic. Patients with ICDs experience some level of anxiety which can impact the number of shocks that they receive from their Device. 100 of these patients will be randomized into one of 2 groups; those receiving three sessions of Cognitive Behavioral Therapy (CBT) and those receiving usual care. We hypothesize that if these ICD patients receive short term (CBT) they will experience less anxiety and have a lower rate of device firings than the patients that did not receive CBT. Furthermore, we will study mechanistic pathways involved in the reduction of anxiety in ICD patients. We will extract initial heart rate variability (HRV) data from device interrogation. We hypothesize that the CBT intervention arm will have a higher normalization of HRV. Patients will repeat questionnaires at 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Currently has an Implantable Cardioverter Defibrillator (ICD)
* Experiences moderate to high anxiety as demonstrated by the the scores on the questionnaires that will be administered

Exclusion Criteria:

* Unwilling to comply with follow-up requirements at 3, 6 and 12 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Patients in the CBT intervention arm will have a higher reduction in anxiety and experience better quality of life compared to usual care at 3 months. | Patients in the CBT arm will have (3) 45min. sessions scheduled over a 3 month period.

SECONDARY OUTCOMES:
Patients in the CBT intervention arm will have a lower rate of firings (shocks). | Patients in both arms will have their ICD's interrogated at 3, 6 and 9 months.

CONTACTS AND LOCATIONS:
Overall Officials: Mina K Chung, MD, Principal Investigator — The Cleveland Clinic; Leopoldo J Pozuelo, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qintar M, George JJ, Panko M, Bea S, Broer KA, St John J, Blissett KA, Ching E, Sears SF, Pedersen SS, Pozuelo L, Chung MK. A prospective study of anxiety in ICD patients with a pilot randomized controlled trial of cognitive behavioral therapy for patients with moderate to severe anxiety. J Interv Card Electrophysiol. 2015 Jun;43(1):65-75. doi: 10.1007/s10840-015-9990-7. Epub 2015 Mar 17. PMID 25779222
- Available data/document: Publication — http://link.springer.com/article/10.1007%2Fs10840-015-9990-7 — A prospective study of anxiety in ICD patients with a pilot randomized controlled trial of cognitive behavioral therapy for patients with moderate to severe anxiety Mohammed Qintar & Jason J. George & Melanie Panko & Scott Bea & Karen A. Broer & Julie St. John & Kecia-Ann Blissett & Elizabeth Ching & Samuel F. Sears & Susanne S. Pedersen & Leopoldo Pozuelo & Mina K. Chung